CLINICAL TRIAL: NCT06675032
Title: Phase I Clinical Trial Protocol of 24-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV24) to Evaluate the Safety and Immunogenicity in Children Aged 2 Months (Minimum 6 Weeks) to 17 Years
Brief Title: Phase I Clinical Trial of PCV24 in Children Aged 2 Months (Minimum 6 Weeks) to 17 Years
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Reinovax Biologics Co.,LTD (Industry)
Collaborators: Shaanxi Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RNCVCT7B001
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- 6~17 years old( PCV24 formulation 1) (Experimental): Dosage form: injection Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 24 months of age-17 years of age: 1 dose.
  Interventions: Biological: PCV24 formulation 1; Biological: Sodium Chloride Injection
- 6~17 years old(PCV24 formulation 2） (Experimental): Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 24 months of age-17 years of age: 1 dose.
  Interventions: Biological: PCV24 formulation 2; Biological: Sodium Chloride Injection
- 24-71 months of age( PCV24 formulation 1) (Experimental): Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 24 months of age-17 years of age: 1 dose.
  Interventions: Biological: PCV24 formulation 1; Biological: Sodium Chloride Injection
- 24-71 months of age(PCV24 formulation 2) (Experimental): Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 24 months of age-17 years of age: 1 dose.
  Interventions: Biological: PCV24 formulation 2; Biological: Sodium Chloride Injection
- 12-23 months of age( PCV24 formulation 1) (Experimental): Dosage form: injection Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 12-23 months age group: 2 doses, at least 2 months apart.
  Interventions: Biological: PCV24 formulation 1; Biological: Sodium Chloride Injection
- 12-23 months of age( PCV24 formulation 2) (Experimental): Dosage form: injection Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 12-23 months age group: 2 doses, at least 2 months apart.
  Interventions: Biological: PCV24 formulation 2; Biological: Sodium Chloride Injection
- 7~11 months of age( PCV24 formulation 1) (Experimental): Dosage form: injection Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 7-11 months age group: 2 doses of primary immunization, with an interval of at least 1 month between the first two doses, and 1 booster dose after 12 months of age.
  Interventions: Biological: PCV24 formulation 1; Biological: Sodium Chloride Injection
- 7~11 months of age(PCV24 formulation 2) (Experimental): Dosage form: injection Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 7-11 months age group: 2 doses of primary immunization, with an interval of at least 1 month between the first two doses, and 1 booster dose after 12 months of age.
  Interventions: Biological: PCV24 formulation 2; Biological: Sodium Chloride Injection
- 2~3 months old (minimum) (6 weeks of age)( PCV24 formulation 1) (Experimental): Dosage form: injection Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 6 weeks to 3 months: one dose at the age of 2, 4 and 6 months for basic immunization, one dose at the age of 12~15 months for booster immunization, and the first dose at the earliest age of 6 weeks.
  Interventions: Biological: PCV24 formulation 1; Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine; Biological: Sodium Chloride Injection
- 2~3 months old (minimum) (6 weeks of age)( PCV24 formulation 2) (Experimental): Dosage form: injection Specification: 0.5 ml/piece Dosage: The preferred part for infants is the anterolateral thigh (vastus lateralis), and the deltoid muscle of the upper arm for toddlers and children, with a dose of 0.5 ml per 1 human use.
  Duration of medication: 6 weeks to 3 months: one dose at the age of 2, 4 and 6 months for basic immunization, one dose at the age of 12~15 months for booster immunization, and the first dose at the earliest age of 6 weeks.
  Interventions: Biological: PCV24 formulation 2; Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine; Biological: Sodium Chloride Injection

INTERVENTIONS:
Biological: PCV24 formulation 1 — 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine formulation 1：Dosage form: Injection Specification:0.5 ml/strip Dosage: The preferred site is the anterolateral thigh (lateral femoral muscle) in infants and the deltoid muscle of the upper arm in infants and children. The preferred dosage for infants is 0.5 ml per dose.
  Dosing schedule:24 months old-17 years old group: 1 dose.12-23 months old group: 2 doses, each dose at least 2 months apart.7-11 months old group: 2 doses of basic immunization, the first two doses at least 1 month apart, and a booster dose after 12 months of age.6 weeks months: 1 dose of basic immunization at each of the ages of 2, 4, and 6 months, and 1 dose of booster immunization at the age of 12-15 months, with the earliest of the first dose at the age of 6 weeks. The first dose is given at 6 weeks of age at the earliest.
  Other Names: 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine
  Arms: 12-23 months of age( PCV24 formulation 1); 24-71 months of age( PCV24 formulation 1); 2~3 months old (minimum) (6 weeks of age)( PCV24 formulation 1); 6~17 years old( PCV24 formulation 1); 7~11 months of age( PCV24 formulation 1)
Biological: PCV24 formulation 2 — 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine formulation 2：Dosage form: Injection Specification:0.5 ml/strip Dosage: The preferred site is the anterolateral thigh (lateral femoral muscle) in infants and the deltoid muscle of the upper arm in infants and children. The preferred dosage for infants is 0.5 ml per dose.
  Dosing schedule:24 months old-17 years old group: 1 dose.12-23 months old group: 2 doses, each dose at least 2 months apart.7-11 months old group: 2 doses of basic immunization, the first two doses at least 1 month apart, and a booster dose after 12 months of age.6 weeks months: 1 dose of basic immunization at each of the ages of 2, 4, and 6 months, and 1 dose of booster immunization at the age of 12-15 months, with the earliest of the first dose at the age of 6 weeks. The first dose is given at 6 weeks of age at the earliest.
  Other Names: 24-Valent Pneumococcal Polysaccharide Conjugate Vaccine
  Arms: 12-23 months of age( PCV24 formulation 2); 24-71 months of age(PCV24 formulation 2); 2~3 months old (minimum) (6 weeks of age)( PCV24 formulation 2); 6~17 years old(PCV24 formulation 2）; 7~11 months of age(PCV24 formulation 2)
Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine — 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine:Dosage form: Injection Specification:0.5 mL/strip Dosage: The preferred site for infants is the anterolateral thigh (lateral femoral muscle), and for toddlers and children, the deltoid muscle of the upper arm.
  Dosing schedule:6 weeks months: 4 doses, one dose each of basic immunization at 2, 4, and 6 months of age, and one dose of booster immunization at 12-15 months of age, with the earliest of the first dose being given at 6 weeks of age. The first dose should be given at 6 weeks of age at the earliest.
  Other Names: Prevenar13®
  Arms: 2~3 months old (minimum) (6 weeks of age)( PCV24 formulation 1); 2~3 months old (minimum) (6 weeks of age)( PCV24 formulation 2)
Biological: Sodium Chloride Injection — Sodium Chloride Injection：Dosage form: Injection Specification:0.5 ml/strip Dosage: The preferred site is the anterolateral thigh (lateral femoral muscle) in infants and the deltoid muscle of the upper arm in infants and children. The preferred dosage for infants is 0.5 ml per dose.
  Dosing schedule:24 months old-17 years old group: 1 dose.12-23 months old group: 2 doses, each dose at least 2 months apart.7-11 months old group: 2 doses of basic immunization, the first two doses at least 1 month apart, and a booster dose after 12 months of age.6 weeks months: 1 dose of basic immunization at each of the ages of 2, 4, and 6 months, and 1 dose of booster immunization at the age of 12-15 months, with the earliest of the first dose at the age of 6 weeks. The first dose is given at 6 weeks of age at the earliest.

SUMMARY:
Phase I clinical trial of 24-valent pneumococcal conjugate vaccine (PCV24) developed by Shanghai Reinovax Biologics Co., LTD will be conducted in children aged 2 Months (Minimum 6 Weeks) to 17 Years . The objective of the study is to evaluate the safety tolerability and immunogenicity of PCV24. The trial is a randomized, blind, controlled combined placebo and positive vaccine control I clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 2~3 months (minimum 6 weeks old) and 7 months old~17 years old, and the guardian of the subject can provide valid identification of the subject and the guardian of the subject.
* Subjects and/or their guardians voluntarily consent to the subjects to participate in this study and sign the informed consent form.
* Subjects and/or their guardians have the ability to understand (non-illiterate) study procedures.
* Female subjects and male subjects of childbearing age agree to use effective contraceptive measures within 6 months from the start of the study to the date of immunization.
* Those who have completed the full course of primary immunization in accordance with the requirements of this clinical trial, and the age before the booster immunization is 12~15 months old, (the interval between the booster immunization time and the last dose of primary immunization is at least 2 months).
* In the opinion of the investigator, the subject's guardian can comply with all the requirements of this clinical trial protocol during the booster phase of the subject.

Exclusion Criteria:

* Individuals who have previously received any type of pneumococcal vaccine or have a history of invasive disease caused by Streptococcus pneumoniae (confirmed by clinical, serological, or microbiological methods).
* Abnormal results from physical examinations or laboratory tests that are deemed clinically significant by a clinician.
* Individuals suspected or diagnosed with fever (axillary temperature ≥37.5℃) within 3 days prior to enrollment; or axillary temperature ≥37.3℃ (for those over 14 years old) or ≥37.5℃ (for those 14 years old or younger) on the day of the first vaccine dose.
* Within 7 days prior to the first dose of vaccination, there is a history of acute illness or acute exacerbation of chronic disease, and systemic application of antibiotics and antiviral medications has been administered; within 3 days prior to the first dose of vaccination, antipyretics, analgesics, and antihistamines (such as acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) have been taken.
* A history of severe allergy to any component of the vaccine being tested, or a history of severe allergy to any vaccine containing tetanus toxoid, or a previous history of severe allergy to any vaccine or medication (including but not limited to: anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrotic reactions, difficulty breathing, angioedema, etc.); or a previous history of severe adverse reactions after the use of any vaccine or medication.
* Subjects who have received inactivated vaccines, subunit vaccines, or recombinant vaccines within 7 days prior to enrollment in the study, or who have received live attenuated vaccines or adenoviral vector vaccines within 14 days prior to enrollment in the study.
* Participants who have received or plan to use any other investigational drug within 3 months prior to the study; those who have received whole blood, plasma, and/or blood products, such as immunoglobulin treatment, within the last 3 months.
* History of thrombocytopenia or other coagulation disorders diagnosed by a hospital, or history of anticoagulant treatment.
* Known to have a current or past history of infectious diseases, such as active tuberculosis, hepatitis B, hepatitis C, and/or human immunodeficiency virus (HIV) infection.
* Known or suspected to have serious chronic diseases, such as liver and kidney diseases, malignant tumors, infections, or allergic skin diseases; or those whose condition is in a progressive stage and cannot be stably controlled.
* Infants under 1 year old with abnormal birth weight (less than 2500 g), or abnormal gestational age (gestational age less than 37 weeks or more than 42 weeks), and those born with abnormal delivery (dystocia, instrumental delivery) or with a history of asphyxia or neurological organ damage.
* Infants under 1 year old have severe eczema or severe jaundice.
* Individuals with severe congenital malformations, developmental disorders, genetic defects, severe malnutrition, or serious chronic diseases (such as Down syndrome, sickle cell anemia, neurological disorders, Guillain-Barré syndrome, etc.).
* Neurological diseases or neurodevelopmental disorders (e.g., febrile seizures, epilepsy, encephalopathy, focal neurological deficits, myelitis or transverse myelitis); history of psychosis or family history.
* History of congenital or acquired immunodeficiency, immunosuppression, or autoimmune diseases, or having received immunomodulatory treatment within the last 6 months, such as immunosuppressive doses of corticosteroids (dose reference: equivalent to prednisone 20 mg/day for more than 7 days); or monoclonal antibodies; or thymosin; or interferons, etc.; but local medications (such as ointments, eye drops, inhalants, or nasal sprays) are allowed.
* Women of childbearing age who are in the breastfeeding period, pregnant, or plan to become pregnant within 6 months after participating in the trial, or have a positive urine pregnancy test result.
* It was learned through inquiry that the subject has no spleen or functional asplenia, as well as any conditions leading to asplenia or splenectomy.
* The subject's guardian may be unable to comply with the study procedures, adhere to agreements, or permanently relocate from the area before the study is completed, or may leave the local area for an extended period during the scheduled visits.
* Researchers believe that any other factors that make the subjects unsuitable for participating in clinical trials may lead to the inability to ensure the maximum benefit for the subjects continuing in the study.
* The subjects received other pneumonia vaccines, apart from the experimental vaccine, before the enhanced immunization.
* The subject has a history of invasive disease caused by pneumococci prior to enhanced immunization (confirmed by clinical, serological, or microbiological methods).
* Researchers believe that if the subjects have any other factors that make them unsuitable for participating in clinical trials, it may lead to the inability to ensure the maximum benefit for the subjects by continuing their participation in the study.
* Persons who have received any type of pneumococcal vaccine prior to enrollment or have a previous history of invasive disease caused by Streptococcus pneumoniae (confirmed by any of the clinical, serologic, or microbiologic methods).
* Abnormal findings on physical examination or laboratory tests that are clinically significant as determined by a clinician.
* Persons with suspected or confirmed fever (axillary temperature ≥37.5°C) within 3 days prior to enrollment; or axillary temperature ≥37.3°C (>14 years of age) or ≥37.5°C (≤14 years of age) prior to (on the day of) the first dose of vaccination.
* History of acute illness or acute exacerbation of chronic illness, systemic treatment with antibiotics and antiviral drugs within 7 days prior to the first dose of vaccination; administration of antipyretic, analgesic, and anti-allergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 3 days prior to the first dose of vaccination.
* A history of severe allergy to any component of the test vaccine or to any vaccine containing tetanus toxoid, or a previous history of severe allergy to any vaccine or medication (including, but not limited to: e.g., anaphylactic shock, anaphylactoid laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, localized anaphylactic necrotic reaction, respiratory distress, angioneurotic edema, etc.); or a previous history of severe side effects to any vaccine or history of severe side effects as described above following drug administration.
* Subjects who have received inactivated, subunit, or recombinant vaccines within 7 days prior to study entry, or live attenuated or adenovirus vector vaccines, etc. within 14 days prior to study entry.
* Those who have received, or plan to use during the study period, any other investigational drug within 3 months prior to enrollment in the study; those who have received whole blood, plasma/ or blood products, such as immunoglobulin therapy within 3 months.
* History of hospital-diagnosed thrombocytopenia or other coagulation disorders or history of anticoagulant therapy.
* Known diagnosis of current/past history of infectious diseases such as: active tuberculosis, hepatitis B, hepatitis C and/or human immunodeficiency virus (HIV) infection.
* Known or suspected serious chronic diseases, such as liver or kidney diseases, malignant tumors, infections, or allergic skin diseases; or if the condition is in a progressive stage that cannot be controlled smoothly.
* Infants less than 1 year of age with abnormal birth weight (<2500 g), or those with abnormal gestational weeks (gestational age <37 or >42 weeks) and births with abnormal labor (obstructed labor, instrumental delivery) or a history of asphyxia or neurological organ damage.
* Infants up to 1 year of age with severe eczema or severe jaundice.
* Suffering from severe congenital malformations or developmental disorders or genetic defects, severe nutritional deficiencies or severe chronic diseases (e.g. Down's syndrome, sickle cell anemia or neurological disorders, Guillain-Barré syndrome, etc.).
* Neurological disorders or neurodevelopmental deficiencies (e.g., febrile convulsions, epilepsy, encephalopathy, focal neurological deficits, encephalomyelitis, or transverse myelitis); history of psychiatric illness or family history.
* History of congenital or acquired immunodeficiency, immunosuppression, or autoimmune disease or treatment with immunomodulators within 6 months, such as immunosuppressive doses of glucocorticoids (dosage reference: equivalent to prednisone 20 mg/day for more than 7 days); or monoclonal antibodies; or thymic peptides; or interferon; but topical medications (e.g., ointments, eye drops, inhalers, or nasal sprays) are allowed.
* Women of childbearing age who are breastfeeding, pregnant, or planning to become pregnant within 6 months of enrollment, or who have a positive urine pregnancy test result.
* Subjects known to be splenic or functionally splenic, and any condition resulting in splenic or splenectomy, upon inquiry.
* Subject guardians may not be able to comply with study procedures, keep appointments, or plan to permanently relocate from the area prior to completion of the study or leave the area for an extended period of time during scheduled visits.
* In the opinion of the investigator, the subject has any other unsuitable factors for participation in the clinical trial that would make continued participation in the study not assured of maximum benefit to the subject.
* Subjects received a pneumonia vaccine other than the experimental vaccine prior to booster immunization.
* Subject has a history of invasive disease caused by Streptococcus pneumoniae prior to booster immunization (confirmed by either clinical, serologic, or microbiologic methods).
* In the opinion of the investigator, the subject has any other unsuitable factors for participation in the clinical trial that would make continued participation in the study not assured of maximum benefit to the subject.

Ages: 6 Weeks to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 2024-04-27 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
2 months ~17 years old incidence of adverse events AE | At the 30 day after every dose vaccination

SECONDARY OUTCOMES:
Incidence of clinically significant abnormality in laboratory examination tests | Day 0 before vaccination and day 4 after vaccination
  12 months ~17 years old:Incidence of clinically significant abnormality in blood routine, blood biochemistry,urine routine and coagulation function test results within 4 days after vaccination
Incidence of serious adverse events (SAE) and | 0-6 months after vaccination
  2 months ~17 years old: incidence of SAEs and AESIs from the first dose of primary immunization to 6 months after full primary immunization.
Incidence of serious adverse events (SAE) | 0-6 months after vaccination
  2 months ~17 years old: incidence of SAEs and AESIs from the first dose of primary immunization to 6 months after full primary immunization.
Proportion of Pneumococcal serotype-specific IgG antibody concentration ≥0.35 μg/ml (seropositive rate) | 30 days after vaccination
  Proportion of IgG antibody concentration ≥0.35 μg/ml
Proportion of Pneumococcal serotype-specific IgG antibody concentration ≥1.0 μg/ml | 30 days after vaccination
  Proportion of IgG antibody concentration ≥1.0 μg/ml
Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) and its growth multiple before immunization | 30 days after vaccination
  IgG GMC 30 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yunong Zhang, Master, Principal Investigator — Shanxi Province Center for Disease Control and Prevention
Locations (1):
- Luzhou District Center for Disease Control and Prevention, Changzhi City, Changzhi, Shanxi, China

IPD SHARING:
Plan to Share IPD: No